CLINICAL TRIAL: NCT02831530
Title: Randomized Short-term Pre-surgical Study to Assess the Effects of Abemaciclib (LY2835219) in Early Breast Cancer Patients
Acronym: ABC-POP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-003425-34; 2015/2288 (Other: CSET Number)
Record Dates: First submitted 2016-07-11; First posted 2016-07-13 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Abemaciclib (Experimental): Patients randomized to the treatment arm will start treatment from 15 days before the surgery (day 1 of the study) to receive the last dose of treatment the day before the surgical procedure (day 14 of the study). Abemaciclib will be taken orally at a dose of 150 mg/ twice a day (Every 12h +/- 2h) on day 1 to day 14. The treatment should be taken in the morning and evening with a big glass of water (250ml) at approximately the same time.
  Interventions: Drug: Abemaciclib
- No treatment (No Intervention)

INTERVENTIONS:
Drug: Abemaciclib
  Arms: Abemaciclib

SUMMARY:
Cyclins CDK4 / 6 are extensively involved in the proliferation and growth of numerous cancers including breast cancer. The objective of this study is to identify if a new preoperative oral treatment, abemaciclib directed against the CDK / 6 compared to no treatment, inhibits tumor growth or induced senescence (aging) tumor.

This early study is offered to women who are going to be operated on for breast cancer with expression of hormone receptor (ER and / or PR). These women will have 3 chances to receive one for up to 14 days in the waiting period of their surgery abemaciclib as tablets. Other patients do not receive treatment. The decision to receive or no treatment will be done by a random computer draw.

The drug's effectiveness will be evaluated primarily on the biological parameters of the tumor itself when comparing surgery to before treatment. These results biomarkers will allow us to better know how this treatment and eventually will be used in future to identify patients for whom treatment with abemaciclib more efficiency.

Patients treated in the protocol will then receive treatment entirely conventional in their breast cancer within the parameters of their tumors: their participation is very limited in time.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Female patients aged 18 years or older.
3. Histologically or cytologically confirmed untreated invasive carcinoma of the breast
4. Candidates for initial breast surgery with a minimum tumor size of 11 mm measured by breast ultrasound. Bilateral and multifocal tumors are allowed, assuming tumor evaluations and pre- and post-treatment biopsies are performed in the same target lesion.
5. HR-positive (defined as either ER and or PR expression >10% by immunohistochemistry or by PCR) irrespective of HER2 status.
6. No evidence of metastatic disease.
7. Eastern Cooperative Oncology Group (ECOG) performance status 0/1.
8. Left ventricular ejection fraction (LVEF) of at least 50%
9. Negative pregnancy test in women of childbearing potential within 14 days prior to treatment initiation (premenopausal or less than 12 months of amenorrhea post-menopause, and who have not undergone surgical sterilization).
10. For women of childbearing potential who are sexually active, agreement to use a highly effective non-hormonal form of contraception or two effective forms of non-hormonal contraception during and for at least 6 months post-treatment.
11. Patients must be affiliated to a social security system

Exclusion Criteria:

1. Patients non-candidate for upfront breast surgery or candidate for neoadjuvant chemotherapy or hormonotherapy.
2. Patients receiving another concomitant anticancer treatment like chemotherapy, immunotherapy, endocrine treatment, or radiotherapy for the currently diagnosed tumor.
3. Known hypersensibility to abemaciclib or any of its components.
4. Difficulty to swallow oral medication.
5. Serious uncontrolled concomitant disease that would put the patient at high risk for treatment-related complications.
6. Patients whose general clinical condition does not consider postponing surgery.
7. Inadequate organ function, evidenced by the following laboratory results:

   * Absolute neutrophil count <1,500 cells/mm3
   * Platelet count <100,000 cells/mm3
   * Hemoglobin <8 g/dL
   * Total bilirubin greater than 1,5 times the upper limit of normal (ULN) (unless the patient has documented Gilbert's syndrome)
   * Aspartate aminotransferase (AST [SGOT]) or alanine aminotransferase (ALT [SGPT]) >3 x ULN
   * Serum creatinine >2 mg/dL and/or clearance creatinine <50mL/min (calculated by Cockcroft-Gault method)
8. Patients with serious preexisting medical conditions that, in the judgment of the investigator, would preclude participation in this study (for example, history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis).
9. Patients with a personal history within the last 12 months of any of the following conditions: syncope of cardiovascular etiology, ventricular tachycardia, ventricular fibrillation, or sudden cardiac arrest.
10. Patients assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.
11. Pregnant or breastfeeding patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2016-03-16 (Actual); Primary Completion 2018-02-02 (Actual); Study Completion 2018-02-02 (Actual)

PRIMARY OUTCOMES:
Anti-proliferative response | Assessed 15 days after randomization
  The primary endpoint is the percentage of patients who at Day 15 have a natural logarithm of percentage positive IHC staining Ki67 of <1 for each study drug (Ki67 "absolute" antiproliferative responders).

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, Val De Marne, France

IPD SHARING:
Plan to Share IPD: No